CLINICAL TRIAL: NCT04981028
Title: The ConNeCT Study: Neurological Complications of Thrombotic Thrombocytopenic Purpura
Brief Title: The ConNeCT Study: Neurological Complications of TTP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 5988
Record Dates: First submitted 2021-07-21; First posted 2021-07-28 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-07

CONDITIONS: Thrombotic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with acute episode of thrombotic thrombocytopenic purpura (TTP): Any adult patients with a suspected diagnosis of TTP (defined by low platelets and anaemia with evidence of red cell breakdown) and confirmed by a low ADAMTS13 enzyme level <10%
  Interventions: Other: Questionnaires (including PHQ-9, TYM and SF-36)
- Healthy volunteers: Non-blood relative / friend / carer
  Interventions: Other: Questionnaires (including PHQ-9, TYM and SF-36)
- Patients with known diagnosis of TTP: Any adult patients with a previously confirmed diagnosis of TTP (more than 12 months ago) based on an ADAMTS13 enzyme level <10% at initial diagnosis
  Interventions: Other: Questionnaires (including PHQ-9, TYM and SF-36)

INTERVENTIONS:
Other: Questionnaires (including PHQ-9, TYM and SF-36) — For the acute group, a questionnaire is completed on neurological symptoms at presentation plus specific questions to include brain imaging performed, treatments received and whether they survived the hospital admission (AQ1). There will be a healthcare practitioner led questionnaire (AQ2) and 3 patient led questionnaires (PHQ-9, TYM and SF-36) plus a supplementary questionnaire (AQ3) completed at 1 week, 1 month, 3 months, 6 months and 12 months following diagnosis. For the chronic TTP group, participants will have a questionnaire completed (CQ1) and 3 patient-led questionnaires (PHQ-9, TYM and SF-36) plus a supplementary questionnaire (CQ2). Where neurological symptoms are present, questionnaires will be completed 6 monthly; where there are no neurological symptoms questionnaires are completed every 12 months. The healthy volunteers will complete participant led questionnaires (namely PHQ-9, TYM, SF-36) plus a supplementary baseline questionnaire at two time points 12 months apart.

SUMMARY:
Thrombotic thrombocytopenic purpura (TTP) is a rare condition, which has a very high risk of death if not recognised and given immediate treatment. TTP is caused by a very low level of an enzyme in the body, called ADAMTS13. A lack of ADAMTS13 causes multiple small clots to form around the body which can disrupt the blood flow to important organs. Although survival has improved significantly, it is now being recognised that patients with TTP may suffer with longer term complications as a result of their condition; literature from the USA reports higher rates of major depression and also poor memory and reduced concentration in patients with TTP. The investigators aim to improve the understanding of the long-term complications and review, for the first time, forward-looking data at multiple time points in patients with TTP in the UK. Both patients with a new diagnosis and patients with a known diagnosis of TTP identified in NHS hospitals will be included, over a minimum duration of 2 years. This will be a questionnaire based study with both doctor led and participant led questionnaires at pre-determined points in time. By improving the understanding and comparing symptoms to that of the general population, the investigators hope to improve the support and tailor the treatments which can be offered to patients with TTP.

ELIGIBILITY:
Inclusion Criteria:

1.Acute episode TTP:

* Adult male or female patient ≥18 years of age at the time of signing the consent form, with a confirmed diagnosis of TTP (initial or relapse) based on ADAMTS13 <10% 2. Known diagnosis of TTP:
* Adult male or female patient ≥ 18 years of age at time of signing the consent form, with a historical confirmed diagnosis of TTP (based on ADAMTS13 at initial presentation <10%) 3. Healthy control:
* Non-blood relative / friend / carer of patients under the care of Haematology clinics at the Royal Liverpool University hospital or other participating centres.

Exclusion Criteria:

1. Acute episode of TTP:

   * Participants less than 18 years old at the time of signing the consent form
   * Patient with ADAMTS13 greater than 10%
   * Patient with cancer or transplant associated MAHA will not be included
   * Patient (or NOK, where patient does not have capacity) not wishing to consent to trial
2. Known diagnosis of TTP:

   * Participants less than 18 years old at the time of signing the consent form
   * Patient with ADAMTS13 greater than 10%
   * Patient with cancer or transplant associated MAHA will not be included
   * Patient (or NOK, where patient does not have capacity) not wishing to consent to trial
3. For healthy control:

   * Participants less than 18 years old at the time of signing the consent form
   * Participant not wishing to consent to trial
   * Any personal or family history of thrombotic microangiopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with thrombotic thrombocytopenic purpura in the United Kingdom
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-06-25 (Actual); Primary Completion 2022-06-25 (Estimated); Study Completion 2022-06-25 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with TTP with neurological complications at acute presentation | 1 week, 1 month, 3 months, 6 months, 12 months
  The primary outcome is to estimate the proportion of both new acute and remission TTP patients developing neurological conditions. These will be reported as counts and percentages with 95% confidence intervals. If we recruit 100 patients in both groups, acute and remission, then we can estimate prevalence rates of 10% with an accuracy of +/- 6%, a 20% prevalence with an accuracy of +/-8% and a 40% prevalence with an accuracy of +/-10%.
The percentage of patients with TTP in remission with long-term neurological complications | 6 months, 12 months, 18 months, 2 years
  The primary outcome is to estimate the proportion of both new acute and remission TTP patients developing neurological conditions. These will be reported as counts and percentages with 95% confidence intervals. If we recruit 100 patients in both groups, acute and remission, then we can estimate prevalence rates of 10% with an accuracy of +/- 6%, a 20% prevalence with an accuracy of +/-8% and a 40% prevalence with an accuracy of +/-10%.

SECONDARY OUTCOMES:
The percentage of 'follow-up' patients with TTP with a depressive disorder, based on PHQ-9 scoring system, compared to the general UK population. | 6 month, 12 months, 18 months, 2 years
  Secondary outcomes include proportion of TTP patients developing depressive or neurological symptoms or having reduced quality of life. These will be reported using counts and percentages, along with 95% confidence intervals. Also, these outcomes will be compared with the corresponding outcomes from the general population (control group). However, as the study is not powered to detect between group differences no formal hypothesis tests will be undertaken and the data will be presented using summary statistics, counts, percentages and 95% confidence intervals.
The percentage of 'follow-up' patients with TTP with neurocognitive deficit, based on TYM scoring system, compared to the general UK population. | 6 month, 12 months, 18 months, 2 years
  Secondary outcomes include proportion of TTP patients developing depressive or neurological symptoms or having reduced quality of life. These will be reported using counts and percentages, along with 95% confidence intervals. Also, these outcomes will be compared with the corresponding outcomes from the general population (control group). However, as the study is not powered to detect between group differences no formal hypothesis tests will be undertaken and the data will be presented using summary statistics, counts, percentages and 95% confidence intervals.
The percentage of 'follow-up' patients with TTP with reduced quality of life, based on SF-36 score, compared to the general UK population. | 6 month, 12 months, 18 months, 2 years
  Secondary outcomes include proportion of TTP patients developing depressive or neurological symptoms or having reduced quality of life. These will be reported using counts and percentages, along with 95% confidence intervals. Also, these outcomes will be compared with the corresponding outcomes from the general population (control group). However, as the study is not powered to detect between group differences no formal hypothesis tests will be undertaken and the data will be presented using summary statistics, counts, percentages and 95% confidence intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Liverpool University Hospital, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided